CLINICAL TRIAL: NCT07077629
Title: Relationship of Scoring Systems With Postoperative Morbidity and Mortality in Geriatric Patients Undergoing Gynecologic Cancer Surgery.
Brief Title: Geriatric Patients Undergoing Gynaecological Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2025-181
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Gynecologic Cancers
Keywords: geriatric surgery; scoring systems; mortality
MeSH Terms: interventions — Morbidity; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric patients undergoing gynecologic cancer surgery: Relationship of scoring systems with postoperative morbidity and mortality in geriatric patients undergoing gynecologic cancer surgery.
  Interventions: Procedure: morbidity and mortality

INTERVENTIONS:
Procedure: morbidity and mortality — Relationship of scoring systems with postoperative morbidity and mortality in geriatric patients undergoing gynecologic cancer surgery.

SUMMARY:
Sınce old age includes variables such as genetics, chronic diseases, lifestyle, aging can be classified as chronological, social, physiological and psychological. According to the World Health Organization's chronological classification, 0-18 years old is considered adolescent, 18-65 years old is young, 65-74 years old is young-old, 74-84 years old is old, and over 85 years old is very old. With advancing age, many physiological changes occur in the body and the risk of non-communicable diseases such as heart and respiratory diseases, cancer, and diabetes increases. Geriatric assessment can be defined as a multidimensional diagnostic process aimed at developing a coordinated and integrated plan for treatment and long-term follow-up in order to determine the medical, psychosocial and functional abilities of an elderly person. Therefore, in order to obtain information about mortality and morbidity in patients undergoing geriatric gynecologic cancer surgery, many risk factors will be evaluated and the usability and reliability of scores and indices will be investigated. For this purpose, many risk scores are used.

DETAILED DESCRIPTION:
Geriatric assessment can be defined as a multidimensional diagnostic process aimed at developing a coordinated and integrated plan for treatment and long-term follow-up in order to determine the medical, psychosocial and functional abilities of an elderly person. Therefore, in order to obtain information about mortality and morbidity in patients undergoing geriatric gynecologic cancer surgery, many risk factors will be evaluated and the usability and reliability of scores and indices will be investigated. For this purpose, many risk scores are used. There are preoperative ASA clinical classification and many postoperative risk protections. ARISCAT risk score is used to investigate postoperative respiratory complications. It consists of a seven-variable model (age, preoperative oxygen saturation (SpO2), respiratory tract infection in the month before surgery, preoperative anemia, surgical incision, duration of surgery and emergency system of the procedure) that separates patients into low, medium and high groups. One of the risk score calculation methods calculated by evaluating comorbidities is the Charlson Comorbidity Index. This score consists of 17 parameters. Participants will be evaluated with the GA-GYN score, which can be separated in this way for geriatric patients and gynecological cancer group surgery. AC surgical risk score is also a score consisting of many parameters such as patients' comorbidities, surgical procedure performed and calculating the risk of disease and death. Walter index will be calculated in order to evaluate these personal 1-year death estimates.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 74 years of age

Exclusion Criteria:

* Incomplete or inadequate patient records

Ages: 74 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: Patients over the age of 74 who underwent gynecological cancer surgery were evaluated retrospectively.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation of Geriatric assesment- Gynaecology( GA-GYN) score with postoperative mortality | postoperative 1 year
  In this score, high scores represent poor results. The GA-GYN score consists of eight parameters:
  1. Need for assistance in taking medications: 1 point
  2. Limited in walking one block : 2 point
  3. Decreased social activity at least sometimes due to physical/emotional health (item from social activity survey):1 point
  4. Number of falls in the last 6 months ≥ 1:3 point
  5. Fair or worse Hearing: 2 point
  6. Age >=72 years: 2 point
  7. Hemoglobin <10 g/dl: 3 point
  8. Creatinine clearance <34 ml/min: 3 point

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vacante M, Cristaldi E, Basile F, Borzi AM, Biondi A. Surgical approach and geriatric evaluation for elderly patients with colorectal cancer. Updates Surg. 2019 Sep;71(3):411-417. doi: 10.1007/s13304-019-00650-3. Epub 2019 Apr 5. PMID 30953329
- [Background] Wozniak SE, Coleman J, Katlic MR. Optimal Preoperative Evaluation and Perioperative Care of the Geriatric Patient: A Surgeon's Perspective. Anesthesiol Clin. 2015 Sep;33(3):481-9. doi: 10.1016/j.anclin.2015.05.012. Epub 2015 Jul 3. PMID 26315633
- [Background] Turrentine FE, Wang H, Simpson VB, Jones RS. Surgical risk factors, morbidity, and mortality in elderly patients. J Am Coll Surg. 2006 Dec;203(6):865-77. doi: 10.1016/j.jamcollsurg.2006.08.026. PMID 17116555